CLINICAL TRIAL: NCT03080012
Title: An Observational Study of Salivary Versus Blood Concentrations of Various Anti-Tuberculosis Drugs in Tuberculosis Patients
Brief Title: Salivary Therapeutic Drug Monitoring of Anti-Tuberculosis Drugs
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan-Willem C Alffenaar, PhD, PharmD, University Medical Center Groningen
Other Study IDs: SALIV-01
Record Dates: First submitted 2017-02-09; First posted 2017-03-15 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Saliva sampling — Stimulated saliva samples are taken using cotton rolls.
Other: Plasma/serum sampling — Simultaneously with saliva sampling.

SUMMARY:
In tuberculosis patients, salivary concentrations will be compared to plasma/serum concentrations of several anti-tuberculosis drugs. If salivary concentrations correctly represent blood concentrations, this non-invasive sampling of saliva could be used for TDM of the tested drugs.

DETAILED DESCRIPTION:
TDM (Therapeutic Drug Monitoring) with blood samples is already part of the treatment of some tuberculosis (TB) patients to reduce development of drug resistance and toxic drug concentrations. Performing TDM with saliva instead of plasma or serum could reduce the burden of blood sampling. This study examines if this non-invasive sampling of saliva could be used for TDM of several anti-TB drugs.

The study is an observational cohort study with adult tuberculosis patients as subjects. The drugs that are studied are isoniazid, rifampicin, ethambutol, pyrazinamide, moxifloxacin, amikacin, kanamycin, capreomycin, ethionamide, prothionamide, cycloserine, terizidone, linezolid, clofazimine, bedaquiline, delamanid, p-aminosalicylic acid (PAS), imipenem-cilastatin, meropenem, ertapenem, amoxicillin-clavulanate and thioacetazone.

Saliva samples will be taken simultaneously with blood samples for standard TDM. Serum/plasma and saliva drug concentrations will be determined with a validated LC-MS/MS (liquid chromatography-tandem mass spectrometry) method. The correlation and linearity between saliva and plasma/serum concentrations will be tested. The saliva-plasma or serum ratio based on area under the time-concentration curve (AUC) is calculated for the investigated anti-TB drugs. Also pharmacokinetic parameters in serum/plasma and saliva will be calculated and compared to provide a complete image of pharmacokinetics of the anti-TB drugs in saliva.

ELIGIBILITY:
Inclusion Criteria:

* Tuberculosis is confirmed by culture or molecular test
* Patient is treated with anti-tuberculosis drugs included in study
* Patient receives Therapeutic Drug Monitoring (TDM) in routine care
* Patient signed informed consent

Exclusion Criteria:

* Patient with severe problems in the oral cavity, making saliva sampling painful

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tuberculosis patients of University Medical Center Groningen Beatrixoord, Haren, The Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Saliva-plasma ratio or saliva-serum ratio | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Ratio of salivary versus blood concentration calculated with salivary and plasma/serum values of area under the time-concentration curve (AUC)

SECONDARY OUTCOMES:
Salivary drug concentration | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Measured drug concentration in saliva
Plasma/serum drug concentration | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Measured drug concentration in plasma or serum
Area under the time-concentration curve (AUC) in saliva and plasma/serum | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Calculated in both saliva and plasma/serum using the drug concentration at all time points.
Peak concentration (Cmax) in saliva and plasma/serum | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Calculated in both saliva and plasma/serum using the drug concentration at all time points.
Time of peak concentration (Tmax) in saliva and plasma/serum | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Calculated in both saliva and plasma/serum using the drug concentration at all time points.
Trough concentration (Cmin) in saliva and plasma/serum | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Calculated in both saliva and plasma/serum using the drug concentration at all time points.
Clearance (Cl) in saliva and plasma/serum | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Calculated in both saliva and plasma/serum using the drug concentration at all time points.
Half-life (t1/2) in saliva and plasma/serum | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Calculated in both saliva and plasma/serum using the drug concentration at all time points.
Elimination constant (Kel) in saliva and plasma/serum | 0, 0.5, 1, 2, 3, 4, 7 hours post-dose for isoniazid, rifampicin, ethambutol and pyrazinamide or 0, 1, 2, 3, 4, 8 hours post-dose for all other drugs
  Calculated in both saliva and plasma/serum using the drug concentration at all time points.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Alffenaar, PhD, PharmD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen (UMCG) Beatrixoord, Haren, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Encoded data can be shared for scientific use up to 15 years after study completion.

REFERENCES:
- [Derived] van den Elsen SHJ, Akkerman OW, Wessels M, Jongedijk EM, Ghimire S, van der Werf TS, Bolhuis MS, Touw DJ, Alffenaar JC. Dose optimisation of first-line tuberculosis drugs using therapeutic drug monitoring in saliva: feasible for rifampicin, not for isoniazid. Eur Respir J. 2020 Oct 22;56(4):2000803. doi: 10.1183/13993003.00803-2020. Print 2020 Oct. No abstract available. PMID 32398308
- [Derived] van den Elsen SHJ, Akkerman OW, Jongedijk EM, Wessels M, Ghimire S, van der Werf TS, Touw DJ, Bolhuis MS, Alffenaar JC. Therapeutic drug monitoring using saliva as matrix: an opportunity for linezolid, but challenge for moxifloxacin. Eur Respir J. 2020 May 7;55(5):1901903. doi: 10.1183/13993003.01903-2019. Print 2020 May. No abstract available. PMID 31980497
- [Derived] van den Elsen SHJ, Akkerman OW, Huisman JR, Touw DJ, van der Werf TS, Bolhuis MS, Alffenaar JC. Lack of penetration of amikacin into saliva of tuberculosis patients. Eur Respir J. 2018 Jan 11;51(1):1702024. doi: 10.1183/13993003.02024-2017. Print 2018 Jan. No abstract available. PMID 29326320